CLINICAL TRIAL: NCT07031544
Title: Efficacy and Influencing Factors of Combined Anterior Limb of Internal Capsule and Nucleus Accumbens Deep Brain Stimulation in Treatment-Refractory Obsessive-Compulsive Disorder
Brief Title: Efficacy and Influencing Factors of ALIC-NAc Deep Brain Stimulation in Treatment-Refractory Obsessive-Compulsive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Huashan Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); Tianjin Anding Hospital (Other); Tianjin Huanhu Hospital (Other); The First Hospital of Hebei Medical University (Other); First Affiliated Hospital of Jinan University (Other); The Second Affiliated Hospital of Xinxiang Medical College (Unknown); the Third Hospital of Mianyang (Unknown)
Responsible Party: Principal Investigator, Zhen Wang, Chief Physician, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMHC-DBS-003
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Obsessive - Compulsive Disorder
Keywords: obsessive-compulsive disorder; deep brain stimulation; anterior limb of internal capsule; nucleus accumbens; activation timing
MeSH Terms: conditions — Compulsive Personality Disorder; Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, randomized, open-label, parallel-group study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- one-month group (Experimental): DBS activation at 30 ± 7 days post-surgery
  Interventions: Device: deep brain stimulation
- two-month group (Experimental): DBS activation at 60 ± 7 days post-surgery
  Interventions: Device: deep brain stimulation
- three-month group (Experimental): DBS activation at 90 ± 7 days post-surgery
  Interventions: Device: deep brain stimulation

INTERVENTIONS:
Device: deep brain stimulation — Deep Brain Stimulation (DBS) involves the use of stereotactic techniques to implant microelectrodes into specific target nuclei within the brain through minimally invasive surgery. These electrodes are connected via leads to a subcutaneously implanted pulse generator, typically placed beneath the clavicle. By delivering low-intensity electrical pulses, DBS suppresses abnormal intracranial neural activity, thereby alleviating symptoms. Long-term stimulation can also induce neuroplastic changes in neural networks and neurotransmitter systems, contributing to the restoration of neurological function.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and influencing factors of the combination of the anterior limb of internal capsule and nucleus accumbens (ALIC-NAc) deep brain stimulation (DBS) in patients with treatment-refractory obsessive-compulsive disorder (OCD). The main questions it aims to answer is:

Does the timing of DBS activation (at 1, 2, or 3 months post-surgery) affect the reduction rate in Y-BOCS scores? Researchers will compare three groups-DBS activated at 1, 2, and 3 months post-surgery-to determine whether earlier or later stimulation leads to greater symptom improvement.

Participants will:

* Undergo surgical implantation of an intracranial neurostimulation system targeting ALIC-NAc
* Be randomly assigned to one of three DBS activation timing groups
* Receive regular clinical assessments over a 6-month follow-up period after activation

DETAILED DESCRIPTION:
This trial adopted a prospective, multicenter, randomized, open-label, parallel-group design. The study population comprised patients with treatment-refractory obsessive-compulsive disorder whose symptoms could not be effectively controlled by pharmacotherapy and psychotherapy. After providing informed consent, participants underwent implantation of an intracranial neurostimulation system, followed by scheduled activation of stimulation post-surgery.

A total of 60 patients were planned for enrollment and randomly assigned to one of three groups based on the timing of stimulation initiation: the one-month group (activation at 30 ± 7 days post-surgery), the two-month group (activation at 60 ± 7 days), and the three-month group (activation at 90 ± 7 days), with 20 participants in each group (1:1:1 allocation). Participants followed the trial schedule for regular assessments. The primary outcome was the difference in Y-BOCS reduction rates among the three groups at 90 ± 7 days after stimulation initiation.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years old;
* a diagnosis of OCD based on The Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5);
* the Y-BOCS total score ≥ 25;
* met the criteria of treatment refractory. Treatment refractory is defined as failed a) Inadequate response or intolerance to at least three adequate trials of selective serotonin reuptake inhibitors (SSRIs), combined with at least two second-generation antipsychotics as augmentation agents.

  b) Inadequate response or intolerance to cognitive behavioral therapy (CBT) consisting of more than 12 sessions conducted concurrently with adequate dosed SSRIs treatment.

Exclusion Criteria:

* Presence of other psychiatric disorders such as organic mental disorders, paranoid personality disorder, or mental retardation.
* Individuals deemed by the investigator to be at significant risk of suicidal behavior based on clinical assessment.
* Presence of severe or unstable cardiovascular, respiratory, hepatic, renal, hematologic, endocrine, neurological, or other systemic diseases.
* History of organic brain disorders, traumatic brain injury, intractable epilepsy, or other neurological conditions.
* Clinically significant abnormalities in physical examination, laboratory tests, electrocardiogram, or imaging during screening or baseline that, in the investigator's judgment, make the individual unsuitable for the study.
* History of implantation of a cochlear implant, cardiac pacemaker, cardiac defibrillator, prior unilateral or bilateral implantation of similar devices, or other surgical procedures within the past six months that may affect study participation as judged by the investigator.
* Contraindications to DBS implantation or deemed unfit for surgery by the investigator.
* Confirmed HIV-positive status.
* Pregnant or breastfeeding women, women of childbearing potential with positive blood/urine HCG results at screening, those unable to use effective contraception during the study, or those planning to conceive within three months after study initiation.
* Participation in another drug or medical device clinical trial currently or within three months prior to screening.
* Any other condition deemed by the investigator to render the individual unsuitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-14 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Obsessive-compulsive symptoms improvement | 3-month after DBS activation
  The severity of OCD symptoms is assessed using the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS). Obsessive-compulsive symptoms improvement is reflected by Y-BOCS reduction rate.

SECONDARY OUTCOMES:
the change scores of CGI score | 1, 2 and 3-month after DBS activation
  The Clinical Global Impressions (CGI) is an invaluable tool for monitoring the treatment outcomes of patients. The CGI actually comprises three companion one-item measures evaluating the following: (a) severity of psychopathology from 1 to 7, (b) change from the initiation of treatment on a similar seven-point scale, and (c) an overall evaluation of the therapeutic effect and side effects.
the change scores of HAMD score | 1, 2 and 3-month after DBS activation
  The Hamilton Depression Rating Scale (HAM-D) is used to quantify the severity of symptoms of depression and is one of the most widely used and accepted instruments for assessing depression. It contains 24 items rated on 5-point scale, with the sum of all items making up the total score, yielding total scores from zero to 96. The higher score means more severity of depression symptoms.
the change scores of HAMA score | 1, 2 and 3-month after DBS activation
  The Hamilton Anxiety Rating Scale (HAM-A) was one of the first rating scales developed to measure the severity of anxiety symptoms. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety and somatic anxiety. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
the change of SF-36 score | 1, 2 and 3-month after DBS activation
  The Short Form-36 Health Survey (SF-36) comprises eight health domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, mental health. It also includes one item assessing perceived health change. These domains can be summarized into two composite scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - the Third Hospital of Mianyang, Mianyang, Sichuan
  - Shanghai Mental Health Center, Shanghai
  - Huashan Hospital, Shanghai
  - Tianjin Huanhu Hospital, Tianjin
  - Tianjin Anding Hospital, Tianjing

REFERENCES:
- [Background] Deuschl G, Herzog J, Kleiner-Fisman G, Kubu C, Lozano AM, Lyons KE, Rodriguez-Oroz MC, Tamma F, Troster AI, Vitek JL, Volkmann J, Voon V. Deep brain stimulation: postoperative issues. Mov Disord. 2006 Jun;21 Suppl 14:S219-37. doi: 10.1002/mds.20957. PMID 16810719
- [Background] Huys D, Kohl S, Baldermann JC, Timmermann L, Sturm V, Visser-Vandewalle V, Kuhn J. Open-label trial of anterior limb of internal capsule-nucleus accumbens deep brain stimulation for obsessive-compulsive disorder: insights gained. J Neurol Neurosurg Psychiatry. 2019 Jul;90(7):805-812. doi: 10.1136/jnnp-2018-318996. Epub 2019 Feb 15. PMID 30770458
- [Background] Denys D, Mantione M, Figee M, van den Munckhof P, Koerselman F, Westenberg H, Bosch A, Schuurman R. Deep brain stimulation of the nucleus accumbens for treatment-refractory obsessive-compulsive disorder. Arch Gen Psychiatry. 2010 Oct;67(10):1061-8. doi: 10.1001/archgenpsychiatry.2010.122. PMID 20921122
- [Background] Belotto-Silva C, Diniz JB, Malavazzi DM, Valerio C, Fossaluza V, Borcato S, Seixas AA, Morelli D, Miguel EC, Shavitt RG. Group cognitive-behavioral therapy versus selective serotonin reuptake inhibitors for obsessive-compulsive disorder: a practical clinical trial. J Anxiety Disord. 2012 Jan;26(1):25-31. doi: 10.1016/j.janxdis.2011.08.008. Epub 2011 Aug 19. PMID 21907540
- [Background] Soomro GM, Altman D, Rajagopal S, Oakley-Browne M. Selective serotonin re-uptake inhibitors (SSRIs) versus placebo for obsessive compulsive disorder (OCD). Cochrane Database Syst Rev. 2008 Jan 23;2008(1):CD001765. doi: 10.1002/14651858.CD001765.pub3. PMID 18253995
- [Background] Huang Y, Wang Y, Wang H, Liu Z, Yu X, Yan J, Yu Y, Kou C, Xu X, Lu J, Wang Z, He S, Xu Y, He Y, Li T, Guo W, Tian H, Xu G, Xu X, Ma Y, Wang L, Wang L, Yan Y, Wang B, Xiao S, Zhou L, Li L, Tan L, Zhang T, Ma C, Li Q, Ding H, Geng H, Jia F, Shi J, Wang S, Zhang N, Du X, Du X, Wu Y. Prevalence of mental disorders in China: a cross-sectional epidemiological study. Lancet Psychiatry. 2019 Mar;6(3):211-224. doi: 10.1016/S2215-0366(18)30511-X. Epub 2019 Feb 18. PMID 30792114
- [Background] Kwon JS, Jang JH, Choi JS, Kang DH. Neuroimaging in obsessive-compulsive disorder. Expert Rev Neurother. 2009 Feb;9(2):255-69. doi: 10.1586/14737175.9.2.255. PMID 19210199
- [Background] Boedhoe PSW, Schmaal L, Abe Y, Alonso P, Ameis SH, Anticevic A, Arnold PD, Batistuzzo MC, Benedetti F, Beucke JC, Bollettini I, Bose A, Brem S, Calvo A, Calvo R, Cheng Y, Cho KIK, Ciullo V, Dallaspezia S, Denys D, Feusner JD, Fitzgerald KD, Fouche JP, Fridgeirsson EA, Gruner P, Hanna GL, Hibar DP, Hoexter MQ, Hu H, Huyser C, Jahanshad N, James A, Kathmann N, Kaufmann C, Koch K, Kwon JS, Lazaro L, Lochner C, Marsh R, Martinez-Zalacain I, Mataix-Cols D, Menchon JM, Minuzzi L, Morer A, Nakamae T, Nakao T, Narayanaswamy JC, Nishida S, Nurmi E, O'Neill J, Piacentini J, Piras F, Piras F, Reddy YCJ, Reess TJ, Sakai Y, Sato JR, Simpson HB, Soreni N, Soriano-Mas C, Spalletta G, Stevens MC, Szeszko PR, Tolin DF, van Wingen GA, Venkatasubramanian G, Walitza S, Wang Z, Yun JY; ENIGMA-OCD Working Group; Thompson PM, Stein DJ, van den Heuvel OA; ENIGMA OCD Working Group. Cortical Abnormalities Associated With Pediatric and Adult Obsessive-Compulsive Disorder: Findings From the ENIGMA Obsessive-Compulsive Disorder Working Group. Am J Psychiatry. 2018 May 1;175(5):453-462. doi: 10.1176/appi.ajp.2017.17050485. Epub 2017 Dec 15. PMID 29377733
- [Background] Thorsen AL, Hagland P, Radua J, Mataix-Cols D, Kvale G, Hansen B, van den Heuvel OA. Emotional Processing in Obsessive-Compulsive Disorder: A Systematic Review and Meta-analysis of 25 Functional Neuroimaging Studies. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Jun;3(6):563-571. doi: 10.1016/j.bpsc.2018.01.009. Epub 2018 Feb 3. PMID 29550459
- [Background] Stein DJ, Costa DLC, Lochner C, Miguel EC, Reddy YCJ, Shavitt RG, van den Heuvel OA, Simpson HB. Obsessive-compulsive disorder. Nat Rev Dis Primers. 2019 Aug 1;5(1):52. doi: 10.1038/s41572-019-0102-3. PMID 31371720